CLINICAL TRIAL: NCT00570219
Title: The Effect of Valproate Treatment on Withdrawal Severity in Benzodiazepine Dependent Opioid Maintenance Treatment Patients
Brief Title: The Effect of Valproate on Benzodiazepine Withdrawal Severity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Helsinki (Other)
Responsible Party: Helena Vorma (principal investigator), Helsinki University Central Hospital, Department of Psychiatry
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PS05BENVAL; KLnro47/2005
Record Dates: First submitted 2007-12-07; First posted 2007-12-10 (Estimated); Last update posted 2008-10-17 (Estimated); Status verified 2008-10

CONDITIONS: Substance Withdrawal Syndrome
MeSH Terms: conditions — Substance Withdrawal Syndrome | interventions — Valproic Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- B (Experimental): Gradual benzodiazepine discontinuation and valproate treatment
  Interventions: Drug: valproate
- A (No Intervention): Gradual benzodiazepine discontinuation

INTERVENTIONS:
Drug: valproate — Valproate 20 mg/kg per day for 2 weeks, reduction during week 3. Conversion of benzodiazepines to an equivalent dose of diazepam (maximum 80 mg per day). Dosage reduced 10 mg daily until 40 mg per day. Reduction then continued 5 mg daily.
  Other Names: Deprakine depot
  Arms: B

SUMMARY:
The aim of this study is to determine whether valproate is effective in the treatment of benzodiazepine withdrawal symptoms in subjects receiving maintenance treatment for opiate dependence.

DETAILED DESCRIPTION:
In Finland, 90% of subjects with opioid dependence are dependent on benzodiazepines too. Concurrent use of opioids and benzodiazepines has increasingly caused deaths.

Benzodiazepine withdrawal treatment usually comprises gradual drug discontinuation. In one study, valproate was shown to improve benzodiazepine discontinuation success in chronic benzodiazepine users. In the present study, the effectiveness of gradual benzodiazepine discontinuation combined with valproate treatment and carried out in an inpatient setting is compared with gradual discontinuation without pharmacological augmentation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of benzodiazepine dependence (DSM IV-R)
* Induction of buprenorphine or methadon maintenance treatment, or need of benzodiazepine withdrawal treatment during ongoing buprenorphine/methadon maintenance

Exclusion Criteria:

* Pregnancy
* History of convulsions
* Unstable somatic diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-02; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
benzodiazepine withdrawal severity | 3 weeks

SECONDARY OUTCOMES:
benzodiazepine use | 4 weeks after treatment
attrition from treatment | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Helena Vorma, MD, Ph.D, Principal Investigator — Deputy chief physician, Helsinki University Central Hospital, Department of Psychiatry; Katila Heikki, Md, Ph.D, Study Director — Chief medical officer, Helsinki University Central Hospital, Department of Psychiatry
Locations (1):
- Helsinki University Central Hospital, Department of Psychiatry, Psychiatric Unit for Drug Dependence, Helsinki, Uusimaa, Finland